CLINICAL TRIAL: NCT06559124
Title: Effect of Kinesio Tape on Pain, Muscle Strength, Functionality and Kinesiophobia in Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, Principal Investigator, University of Beykent
Allocation: Not Applicable | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UBeykent-10
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-08

CONDITIONS: Physiotherapy; Kinesiotaping
Keywords: Impingement syndrome; functionality; kinesiophobia
MeSH Terms: conditions — Kinesiophobia | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: After giving the necessary verbal and written information about the study, patients with informed consent will be randomized and divided into 3 groups of 20 people each. The randomization and treatment of the cases will be done by the same researchers. The evaluation will be carried out before and after the treatment by another researcher who is blind to which group the participants are in.
  After the initial evaluations are completed, Group 1 will receive 15 sessions of traditional physiotherapy + placebo kinesiotape every day for 3 weeks. In the 2nd group, kinesiotape will be applied with traditional physiotherapy + facilitation method. In the third group, kinesiotape will be applied with traditional physiotherapy + inhibition method.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Grup A: Traditional Physiotherapy + Sham Kinesiotape (Sham Comparator): Traditional Physiotherapy: A total of 15 sessions of joint range of motion, stretching exercises and strengthening exercises will be applied 5 days a week for 3 weeks, each session lasting 45 minutes. Friction massage will be applied. In addition, ultrasound, TENS and cold packs will be applied to the patients according to their tolerance.
  Sham Kinesiotape: 2 days a week, 6 times in total, following conventional physiotherapy for 3 weeks. Kinesio tape 10 cm I strips will be applied on the acromioclavicular joint in the sagittal plane and in the transverse plane from the distal deltoid without applying tension. The tape will be applied twice a week in total, remaining for 3 days and released one day after each application.
  Interventions: Other: Traditional Physiotherapy + Sham Kinesiotape
- Grup B: Kinesiotape with Facilitation Method + Traditional Physiotherapy (Experimental): In addition to traditional physiotherapy, traditional physiotherapy will be applied 2 days a week, 6 times in total, followed by 3 weeks. Kinesio tape has been developed to reflect the properties of the skin, its thickness is similar to the epidermis layer of the skin, and its elasticity is similar to the elastic properties of human skin. Participants should be informed that the patch will remain for several days and will not be removed by bathing or swimming. Kinesio tape will be applied to the deltoid muscle with the starting point at 0 tension while the arm is in a relaxed position and will be slightly heated. It will be applied in addition to traditional physiotherapy 2 days a week for 3 weeks.
  Interventions: Other: Kinesiotape with Facilitation Method + Traditional Physiotherapy
- Grup C: Kinesiotape with Inhibition Method + Traditional Physiotherapy (Experimental): In addition to traditional physiotherapy, traditional physiotherapy will be applied 2 days a week, 6 times in total, followed by 3 weeks.
  Kinesio tape will be applied to the deltoid muscle with inhibition and mechanical correction technique, and to the supraspinatus muscle with inhibition technique twice a week, 3 days apart. First of all, it will be applied to the deltoid muscle with the inhibition technique. Y-shaped kinesio tape will be placed 3 cm below the humerus tuberculum deltoidea without stretching. During application, the shoulder will be in maximum extension and external rotation for the front arm of the Y strip, and in 45 degrees transverse flexion and horizontal adduction for the rear arm of the Y strip.
  Interventions: Other: Kinesiotape with Inhibition Method + Traditional Physiotherapy

INTERVENTIONS:
Other: Traditional Physiotherapy + Sham Kinesiotape — As exercise training, joint range of motion, flexion and abduction external cycle will be practiced with the gymnasts.
  Circumference measurements will be taken for shoulder bone swelling and for atrophy.
  Shoulder joint mobilizations will be applied (posterior cutting for flexion limitation, downward shifting and scapular mobilizations for abduction limitation).
  Flexion and abduction will be stretched externally. Friction massage will be applied. Strengthening exercises for flexion, abduction and external rotation in the lower and upper segments of the shoulder with dumbbells and theraband, shoulder wheel and finger ladder will be practiced.
  Codman exercises and staff exercises will be practiced.
  Arms: Grup A: Traditional Physiotherapy + Sham Kinesiotape
Other: Kinesiotape with Facilitation Method + Traditional Physiotherapy — Kinesio tape will be applied with 0 tension at the starting point when the arm is in a relaxed position and will be slightly heated. Since the deltoid muscle is a three-headed muscle, it will be applied with 0 tension in the flexed position at the elbow, for the front part, the arm with the elbow in full extension, and for the middle part of the deltoid, the I tape will be applied along the muscle without applying tension.
  Arms: Grup B: Kinesiotape with Facilitation Method + Traditional Physiotherapy
Other: Kinesiotape with Inhibition Method + Traditional Physiotherapy — The Y-shaped kinesio tape will be placed on the deltoid muscle with inhibition and mechanical correction technique, and the Y-shaped kinesio tape will be placed on the supraspinatus muscle with inhibition technique, 3 cm below the humerus tuberculum deltoidea without tension. The Y tape will be applied along the outer edge of the anterior deltoid of the forearm with 15-25% light tension, and the posterior arm will be applied along the outer edge of the posterior deltoid with 15-25% light tension up to the lateral acromion. The last 3-5 cm of the tails will be applied to their permanent locations without tension. The shoulder will be held in maximum transverse extension and external rotation for the forearm of the Y support, and in 45 degrees transverse flexion and horizontal adduction for the posterior arm of the Y support. In addition, ultrasound, electrotherapy and cold application will be applied to the participants depending on their tolerance.
  Arms: Grup C: Kinesiotape with Inhibition Method + Traditional Physiotherapy

SUMMARY:
The aim of the study is to compare the effects of different kinesiotape applications in addition to traditional physiotherapy on shoulder pain, joint range of motion, muscle strength, functionality and kinesiophobia in patients diagnosed with shoulder impingement syndrome within and between groups.

Subacromial space; At the bottom, it is the region limited by the humeral head and tuberculum major, acromion (anterior 1/3 of the acromion), coracoacromial ligament, coracoid process and acromioclavicular joint and acromioclavicular ligament. The rotator cuff muscles pass through this area and move within it. In anteroposterior radiographs taken with the shoulder in 0° abduction, the distance between the acromion and the humeral head is approximately 1.1 cm (1.0-1.5 cm). Between these two structures are the rotator cuff (mostly the supraspinatus tendon), the long head of the biceps muscle, the bursa, and the coracoacromial ligament.

When incompatibility is observed between the mentioned bone structures, it causes pressure on the subacromial structures. Subacromial impingement syndrome is one of the most common causes of shoulder pain. The complaint of the majority of patients is pain radiating to the shoulder and arm, especially during overhead movements.

Examples of overhead activities in these people include hanging curtains, reaching on a shelf, combing hair, or lifting an object. Subacromial impingement syndrome is a complex disease that occurs not only as a result of compression of the rotator cuff muscles under the acromion, but also due to a combination of external and internal causes. While the diagnosis of the disease can be made with a good history and physical examination, the diagnosis must also be supported by imaging methods.

DETAILED DESCRIPTION:
When applied to the skin and muscle, kinesiology tape affects the mechanoreceptors sensitive to tension, loading, pressure and shear forces by changing the length of the skin and superficial fascia and the tension of the muscle fibers.

This can lead to significant changes in muscle movement and tone. In particular, slow pressure stimulation on connective tissue alters the effect on mechanoreceptors and may affect gamma motor neuron firing and muscle tone regulation. Kinesio tape can be effective in increasing proprioceptive ability, especially in the middle of movement. In this range, muscle receptors are active while ligament mechanoreceptors are inactive. Understanding joint movement and position can be effective in improving proprioception by stimulating sensory afferent transmission.

Inhibition techniques are divided into two; Autogenic and reciprocal inhibition. It occurs when the contraction of certain muscles is inhibited due to activation of the Golgi tendon and muscle spindle. These two myotendinous proprioceptors, located in and around joints and muscles, help manage muscle control and coordination by responding to changes in muscle tension and length.

Although there are studies in the literature on traditional physiotherapy and kinesio taping in patients with shoulder impingement syndrome, no study has been found that includes different kinesio taping techniques and all evaluation parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with subacromial impingement syndrome,
* Between the ages of 45-65, without a history of shoulder injury other than subacromial impingement and/or shoulder symptoms requiring treatment for the last 1 year,
* Those who have not had any shoulder surgery before,
* Patients who agree to participate in the study will be included in the study.

Exclusion Criteria:

* Those who do not meet the inclusion criteria and have a history of shoulder fracture, dislocation and/or cervical radiculopathy,
* Presence of frozen shoulder, previous shoulder surgery,
* Having received local corticosteroid injection/treatment to the shoulder joint in the last 3 months,
* Presence of neuromuscular disease, pregnancy,
* Those with a history of cancer, unstable angina, systemic inflammatory joint disease,
* Situations where exercise is contraindicated,
* Patients with orthopedic, rheumatic or congenital disease in the affected upper extremity and communication problems will be excluded from the study.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Visuel Analog Scale (VAS) | 3 weeks
  Visuel analog scale is a scale where the intensity of pain is marked on a 10 cm horizontal/vertical line. The point "0" indicates no pain, and the point "10" indicates maximum pain. Participants will be asked to mark the point that represents their pain at the beginning and after treatment. The marked point will then be measured with a ruler and recorded in "cm". A higher value indicates more pain. The reliability of the assessment is r=0.79 and the retest validity is r=0.97.
Joint Range of Motion (ROM) | 3 weeks
  It refers to the measurement of the amount of movement around a particular joint. This measurement is usually made during a physical therapy evaluation. Physiotherapists measure joint range of motion with the help of a tool called a goniometer. The midpoint of the digital goniometer will be fixed by holding it with the hand, with the pivot point for movement of the shoulder joint placed on the greater tubercle of the humerus bone. A digital goniometer will be used to measure shoulder joint range of motion.
Muscle Strength | 3 weeks
  The maximal power that can be generated by a specific muscle or muscle group. Muscular strength is the ability of the muscle to resist resistance. In assessing muscle strength, the force or torque applied during maximal voluntary contraction is measured. Evaluation is performed to detect peripheral muscle weakness before treatment, to plan a personalized resistance exercise training program, and to evaluate post-treatment effectiveness. Many methods including voluntary and involuntary contractions are used to measure muscle strength. The physiotherapist who will perform the application must choose the correct, sensitive and most reliable test appropriate to the clinical conditions.
Disabilities of the Arm, Shoulder and Hand (DASH) | 3 weeks
  The questionnaire, which evaluates upper extremity functions and gives an idea about upper extremity functionality, consists of 3 parts: symptoms and daily living activities, sports and musician module. The questionnaire consists of 30 items assessing symptoms and activities of daily living. 21 questions in the survey evaluate difficulty in daily life activities, 5 questions evaluate body symptoms (pain, weakness, stiffness, numbness), and the remaining 4 questions evaluate work skills, sleep status, social function and the patient's self-confidence. A 5-grade system is used in scoring the survey. In the scoring scale from 1 to 5, 1 means "no difficulty" and 5 means "I cannot do it at all".
  The time to complete the survey is 5-7 minutes and it is a survey that patients can easily answer on their own. The highest score is 100, and high scores indicate low patient functionality.
Tampa Kinesiophobia Scale (TKS) | 3 weeks
  The level of kinesiophobia will be assessed with the Tampa Kinesiophobia Scale (TKS). The scale consists of 17 questions. The scoring varies between 17-68, with higher scores indicating higher kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin ŞAHBAZ, Lecturer, Principal Investigator — Beykent University
Locations (1):
- Yasemin ŞAHBAZ, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poppen NK, Walker PS. Forces at the glenohumeral joint in abduction. Clin Orthop Relat Res. 1978 Sep;(135):165-70. PMID 709928
- [Background] Neer CS 2nd. Anterior acromioplasty for the chronic impingement syndrome in the shoulder: a preliminary report. J Bone Joint Surg Am. 1972 Jan;54(1):41-50. No abstract available. PMID 5054450
- [Background] Neer CS 2nd. Impingement lesions. Clin Orthop Relat Res. 1983 Mar;(173):70-7. No abstract available. PMID 6825348
- [Background] Winter JA, Allen TJ, Proske U. Muscle spindle signals combine with the sense of effort to indicate limb position. J Physiol. 2005 Nov 1;568(Pt 3):1035-46. doi: 10.1113/jphysiol.2005.092619. Epub 2005 Aug 18. PMID 16109730
- [Background] Visscher CM, Ohrbach R, van Wijk AJ, Wilkosz M, Naeije M. The Tampa Scale for Kinesiophobia for Temporomandibular Disorders (TSK-TMD). Pain. 2010 Sep;150(3):492-500. doi: 10.1016/j.pain.2010.06.002. Epub 2010 Jul 3. PMID 20598804